CLINICAL TRIAL: NCT01894035
Title: Study to Assess the Compliance of Patients With Pulmonary Arterial Hypertension Treated With Inhaled Iloprost.
Brief Title: Non-interventional Multi-center Study on Patients Under Routine Treatment of Pulmonary Arterial Hypertension (PAH) With Inhaled Iloprost Using I-Neb as a Device for Inhalation
Acronym: COMPHI
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16755; VE1310PT (Other: Company internal)
Record Dates: First submitted 2013-07-03; First posted 2013-07-09 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Ventavis; Patient compliance
MeSH Terms: conditions — Hypertension, Pulmonary; Patient Compliance | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Iloprost (Ventavis, BAYQ 6256)

INTERVENTIONS:
Drug: Iloprost (Ventavis, BAYQ 6256) — Patients Diagnosed with Pulmonary Arterial Hypertension, Functional Class NYHA/WHO III, for whom was prescribed inhaled Iloprost.

SUMMARY:
This pilot, non-interventional, company-sponsored, multi-center study documents observational data on patients under routine treatment of Pulmonary Arterial Hypertension (PAH) with inhaled iloprost (using I-Neb device for the inhalation).

The planned study recruitment time is 18 months. The maximum follow up period in this study will be 12 months.

The data will be collected from patients who have initiated the treatment mentioned above (inhaled iloprost using I-Neb device) since February 1st, 2013.

Frequency of visits and procedures will be performed under routine conditions. The primary objective of this study is to assess the compliance of patients with WHO/NYHA (World Health Organization/New York Heart Association) functional Class III Pulmonary Arterial Hypertension treated with Inhaled Iloprost in clinical practice, using the I-neb Insight tool.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18years old), male or female
* Diagnosis of Pulmonary Arterial Hypertension, Group I of the Dana Point Pulmonary Hypertension classification (Diagnosis made at the discretion of the attending investigator, including mPAP ≥ 25 mmHg at rest, as measured by right heart catheterization.)
* The treating physician has chosen to initiate the treatment with inhaled iloprost with I-Neb device for the application, as described in the Summary of Product characteristics (SmPC).
* WHO/NYHA functional class III
* Willing to participate in the study (Informed Consent Sign)
* Patients who received the first inhaled iloprost treatment with I-Neb from February 1st, 2013.

Exclusion Criteria:

* Any contraindication for the treatment with Ventavis as described in the Summary of Product characteristics (SmPC)
* Patients are not to be enrolled if they were treated with inhaled iloprost with I-Neb or any other device for the application in the past, before the start of the observation period (February 1st, 2013)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Diagnosed with Pulmonary Arterial Hypertension, Functional Class NYHA/WHO III, for whom the treating physician has chosen to initiate the treatment with inhaled iloprost using I-Neb as the device for inhalation since 1st of February of 2013.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Percentage of compliant patients | Up to 12 months
  The compliance will be assessed by the mean daily number of Inhalations and mean daily dose of Ventavis at around months 6 and 12 for each patient (Data will be collected via the I-neb Insight). For this observational study, a patient is considered compliant if the mean daily number of inhalations and mean daily dose are within 80 to 120% of prescribed. Otherwise, the patient will be considered as non-compliant.

SECONDARY OUTCOMES:
Observed treatment duration days | Up to 12 months
Expected treatment duration days | Up to 12 months
Changes in WHO/ NYHA Functional Class | Up to 12 months
Change in 6 MWDT (6 minute walking distance test) scale value | Up to 12 months
Change in Dyspnea Borg CR (category ratio) 10 scale value | Up to 12 months
Quality of life using validated scales (EuroQol questionnaire [EQ-5D], Living with Pulmonary Hypertension questionnaire [LPH]) | Up to 12 months
Adjusted percentage treatment duration | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Portugal